CLINICAL TRIAL: NCT01684839
Title: Treatment of Painful Digital Neuroma Using A Pedicled Nerve Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other); The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB-TS-120127; TSCHEN411206 (Other: Ethics Committee of HeBei Province)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2012-06

CONDITIONS: Painful Digital Neuroma
Keywords: Painful digital neuroma; nerve defect; dorsal branch of the digital nerve; digital nerve; pedicled nerve flap; Pain Disorder Associated with Psychological and Physical Factors
MeSH Terms: interventions — Surgical Flaps

ARMS (1):
- new surgical treatment (Other): Treatment of Painful Digital Neuroma Using A Pedicled Nerve Flap taken from the homolateral dorsal branch of the digital nerve.
  Interventions: Device: Pedicled nerve flap

INTERVENTIONS:
Device: Pedicled nerve flap — This nerve flap is a vascularized nerve graft
  Other Names: Surgical flap; Island flap

SUMMARY:
Neuroma excision and digital nerve reconstruction remain the best option for the treatment of Painful Digital Neuroma (PDN). When the distal nerve end is preserved, conventional nonvascularized nerve grafting is the primary option to bridge the defect. The investigators hypothesize the pedicled nerve flap taken from the dorsal branch of the homolateral digital nerve is better than conventional methods for reconstruction of the digital nerve defect after painful neuroma resection.

This study reports treatment of painful digital neuroma using a pedicled nerve flap taken from the dorsal branch of homolateral digital nerve. From May 2007 to March 2010, the patients had previous nerve injuries with or without nerve repair. The mechanisms of injury include sharp cut, avulsion and crush. The defects were between the middle of the distal phalanx and the palmar digital crease.

DETAILED DESCRIPTION:
Our selection criteria in this study included a patient with PDN in a scarred wound bed or poor coverage, a PDN located between the middle of the distal phalanx and the palmar digital crease, and a defect of the digital nerve after neuroma resection equal to or less than 3 cm in length. The exclusion criteria included a PDN in healthy soft tissue, a digital nerve defect longer than 3 cm, injury to the course of the pedicle or the donor nerve, and a thumb neuroma. A finger with a small distal end of the digital nerve was also excluded, because neurorrhaphy was extremely difficult in this situation.

ELIGIBILITY:
Inclusion Criteria:

* a patient with PDN in a scarred wound bed or poor coverage
* a PDN located between the middle of the distal phalanx and the palmar digital crease
* a defect of the digital nerve after neuroma resection equal to or less than 3 cm in length

Exclusion Criteria:

* a PDN in healthy soft tissue
* a digital nerve defect longer than 3 cm
* injury to the course of the pedicle or the donor nerve
* a thumb neuroma

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD., Study Chair — The Second Hospital of Tangshan
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Herndon JH, Eaton RG, Littler JW. Management of painful neuromas in the hand. J Bone Joint Surg Am. 1976 Apr;58(3):369-73. PMID 1262369
- [Result] Tupper JW, Booth DM. Treatment of painful neuromas of sensory nerves in the hand: a comparison of traditional and newer methods. J Hand Surg Am. 1976 Sep;1(2):144-51. doi: 10.1016/s0363-5023(76)80008-1. PMID 1032972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine patients were included in the study. These patients were treated with the pedicled nerve flap. The type of location was medical clinic.
Pre-assignment Details: No wash out, run-in or transition happened in the study.
Period: Overall Study
Arm/Group | New Surgical Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | New Surgical Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Region of Enrollment [Number; unit: participants]
  China | 9

OUTCOME MEASURES:

1. Primary Outcome: Static 2-point Discrimination Test
Description: The Static 2-point Discrimination Test determined the minimal distance at which a subject can sense the presence of two needles. The modified American Society for Surgery of the Hand guidelines was used to stratify the 2PD measurements (excellent <6 mm; good 6-10 mm; fair 11-15 mm; poor >15 mm). The test points were at the center of the radial or ulnar portion of the finger pulp (i.e., injury side). Each area was tested 3 times with a discriminator (Ali Med, Dedham, MA). Two out of 3 correct answers were considered proof of perception before proceeding to another lower value. We stopped at 4mm as a limit of 2PD and consider this normal. The measurements were performed at a single time point at the final follow up.
Time Frame: 20-26 months postoperatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | New Surgical Treatment
Number analyzed (Participants) | 9
mm | 7.3 (2.0)

2. Secondary Outcome: Cold Intolerance Severity Score (CISS) Questionnaire
Description: The maximum score was 100 and was grouped into 4 ranges (0-25; 26-50; 51-75; and 76-100), corresponding to mild, moderate, severe, and extreme severity, respectively.
Time Frame: 20-26 months postoperatively
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Tinel's Sign
Description: Tinel's sign was graded as the following: grade 1=none; grade 2=mild, slight tingle; grade 3=moderate, very uncomfortable; and grade 4=severe, patient unable to use hand because of any stimulation of the neuroma
Time Frame: 20-26 months postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | New Surgical Treatment
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes